CLINICAL TRIAL: NCT05305560
Title: A Multicentre Randomised, Double-Blind, Placebo-controlled, Study to Evaluate the efficAcy and Safety of Oral IVErmectin Tablets in the Prevention of COVID-19
Brief Title: A Study to Evaluate the Efficacy and Safety of Ivermectin in COVID-19 Prevention
Acronym: SAIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedinCell S.A (Industry)
Collaborators: Violaine Desort-Hénin, DVM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mdc-TTG-CT-002; 2021-001938-19 (EudraCT Number)
Record Dates: First submitted 2022-03-28; First posted 2022-03-31 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: Prophylaxis; RT-PCR test
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active IMP (Experimental)
  Interventions: Drug: Ivermectin Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo tablets

INTERVENTIONS:
Drug: Ivermectin Tablets — Daily ivermectin tablets intake for 28 days ; 200 mcg/kg on D1 then 100 mcg/kg daily from D2 to D28.
  Arms: Active IMP
Drug: Matching placebo tablets — Daily placebo tablets intake for 28 days
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, study to evaluate the efficacy and safety of oral ivermectin tablets versus placebo for COVID-19 prophylaxis

DETAILED DESCRIPTION:
This trial comprises a total observation period of up to 56 days (an on-treatment period of up to 28 days and a safety follow-up of up to 28 days).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years, inclusive.
2. Body weight >45 kg.
3. Body Mass Index >18.5.
4. Close contact with a person who has a PCR-confirmed SARS-CoV-2 infection within 5 days before screening.
5. Only one member in the same household will be enrolled.
6. Participants must be able to give informed consent and comply with the study's scheduled events/visits and study assessments.
7. SARS-CoV-2 positive index case must be able to give consent to enable collection of the documented positive PCR test.
8. Female participants of childbearing potential must use a highly effective method of contraception for the duration of the trial.

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Participants who have been administered COVID-19 vaccine prior to the inclusion or have a planned vaccination during the duration of the study.
3. A positive COVID-19 result (PCR or antigen test) within 8 days of screening.
4. Presence of typical COVID-19 symptoms (fever >38°C, SpO2 below 93%, dyspnoea, difficulty breathing, chills, repeated shaking with chills, ageusia, anosmia, cough, myalgia, headache) in the past 48 hours prior to screening.
5. Hypersensitivity to any component of ivermectin.
6. Participants who have been administered ivermectin within 30 days prior to screening.
7. Participation in another interventional trial within the last 30 days or 5 half-lives of the IMP of the other trial, whichever comes first.
8. Participants with gastrointestinal erosions and ulcers (e.g. erosive esophagitis, stomach ulcers, ulcerative colitis etc.).
9. History of neurotoxicity with ivermectin or other para-glycoprotein (p-gp) substrates or inhibitors.
10. Current use of monoclonal antibodies for the treatment of COVID-19.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kostova, MD, Principal Investigator — Medical Center Medic Ltd.
Locations (1):
- Medical Center Medic Ltd., Sofia, Bulgaria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active IMP | Placebo
Started | 200 | 199 (1 participant on placebo did not receive treatment as no kit was available on site)
Completed | 200 | 199
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active IMP | Placebo | Total
Number analyzed (Participants) | 200 | 199 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.86 (11.84) | 39.99 (12.03) | 40.42 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant who was randomized to placebo did not receive treatment as the IMP Kit was not available at the site. They were not included in the analyses
  Participants
    Female | 81 | 90 | 171
    Male | 119 | 109 | 228
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bulgaria | 200 | 199 | 399

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Prophylaxis
Description: Number of laboratory-confirmed COVID-19 infections in each group between baseline and Day 28
Time Frame: From Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Active IMP | Placebo
Number analyzed (Participants) | 200 | 199
Participants | 30 | 105

2. Secondary Outcome: COVID-19 Symptoms Development
Description: Number of symptomatic Participants according to the WHO COVID-18 scale
Time Frame: From Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Active IMP | Placebo
Number analyzed (Participants) | 200 | 199
Participants | 28 | 97

3. Secondary Outcome: COVID-19 Prophylaxis Timeframe
Description: Time to change from baseline in negative RT-PCR to positive RT-PCR
Time Frame: From Day 1 to Day 28
Population: Participants who've had a positive RT-PCR during the trial
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active IMP | Placebo
Number analyzed (Participants) | 30 | 105
days | 9 (1.39) | 8.10 (2.14)

4. Secondary Outcome: COVID-19 Hospitalisations
Description: Proportion of COVID-19 related hospitalisations
Time Frame: From Day 1 to Day 56
Population: Partcipants who had COVID-19 related hospitalisatoin episodes
Measure: Number; unit: participants
Arm/Group | Active IMP | Placebo
Number analyzed (Participants) | 200 | 199
participants | 0 | 0

5. Secondary Outcome: COVID-19 Mortality
Description: Proportion of COVID-19 related mortality
Time Frame: From Day 1 to Day 56
Population: Participants who suffered a COVID-19 related death
Measure: Number; unit: participants
Arm/Group | Active IMP | Placebo
Number analyzed (Participants) | 200 | 199
participants | 0 | 0

6. Secondary Outcome: To Assess the Safety and Tolerability of IVM Given for a Period of 28 Days
Description: Descriptive comparison of AE rates and severity/seriousness between IVM and placebo
Time Frame: 56 days
Population: All participants who have received at least a single dose of the allocated treatment
Measure: Number; unit: participants
Arm/Group | Active IMP | Placebo
Number analyzed (Participants) | 200 | 199
participants
  Adverse events | 49 | 109
  Serious adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 days
Description: Adverse events were collected passively upon Participant declaration.
Arm/Group | Active IMP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/199
Other Adverse Events (participants affected / at risk) | 49/200 | 109/199
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active IMP (N=200) | Placebo (N=199)
COVID-19 (Infections and infestations) | 30 (30) | 109 (109)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Vertigp (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Basophil count increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can present and discuss the results but publication is subject to the sponsor's prior approval

DOCUMENTS (2):
  • Study Protocol (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT05305560/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05305560/SAP_001.pdf